CLINICAL TRIAL: NCT01769300
Title: Improving the Medication Management of Patients With Attention-Deficit Hyperactivity Disorder
Acronym: ePROS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: American Academy of Pediatrics (Other)
Collaborators: University of Colorado, Denver (Other); QED Clinical, Inc (Unknown); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: UB5MC20286
Record Dates: First submitted 2013-01-11; First posted 2013-01-16 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Attention Deficit-hyperactivity Disorder
Keywords: Clinical decision support; Electronic health records; Electronic medical records; Attention deficit-hyperactivity disorder; Primary care Pediatric research network
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control practices (No Intervention): Practices that do not use the ADHD clinical decision support
- Clinical decision support (Experimental): Electronic health record-based clinical decision support for ADHD medication titration.
  Interventions: Behavioral: Clinical decision support for medication titration

INTERVENTIONS:
Behavioral: Clinical decision support for medication titration — Electronic health record-based clinical decision support for ADHD medication titration.
  Arms: Clinical decision support

SUMMARY:
The specific aim of this cluster-randomized (site) comparative effectiveness research study is to determine whether children who are (1) 5-12 years of age, (2) cared for in ePROS practices or clinics using an electronic health record (EHR), (3) have attention-deficit hyperactivity disorder (ADHD), and (4) are to receive treatment with stimulant medication for the first time in these practices, have superior clinical outcomes if their clinicians have access to an EHR-guided clinical decision support system (intervention group) than if their clinicians have no such access (control group).

DETAILED DESCRIPTION:
In this cluster (site)-randomized trial of clinical decision support for ADHD medication titration, clinicians caring for children with ADHD whose families are initiating stimulant medication at that practice will be followed.

Two groups will be compared; an intervention group, which will receive the intervention-the clinical decision support (CDS)--, and a control group, who will not receive CDS. Over a 6-month period, the CDS will support guideline-based medication titration to achieve optimal symptom control with minimal side effects. The study will track the care delivered to affected children by the practitioners and will assess the endpoints of symptom reduction and side effects. There will also be a sub-study within the larger study which will give the team a better understanding about the pros and cons of consenting parents over the phone.

ELIGIBILITY:
Practice Eligibility Criteria

* Willing to offer the possibility of study enrollment to their patients who have ADHD
* Willing to use the Vanderbilt Assessment Rating Scale to assess and potentially, to monitor ADHD for study subjects
* Utilize Integrated Health Connect as a means to collect the Vanderbilt Assessment Rating Scale
* Use point-of-care reports for subjects enrolled in the study.

Patient Eligibility Criteria

* The child must be between the ages of 5-12 years old
* The child must be starting stimulant medication for the first time
* Parent must be able to speak and read English
* The child must not be diagnosed with a current manic episode, a psychotic disorder, or a pervasive developmental disorder (e.g. autism, Asperger's, Rett's disorder)
* The child must not have reported suicidality or have conduct disorder, per parent/guardian report

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Improvement in symptoms, as measured by the parent-reported Vanderbilt Assessment Scale. | 4 & 6 months after enrollment
  This intervention study tests a clinical decision support system for ADHD treatment.

SECONDARY OUTCOMES:
Side effects as reported on the ADHD Vanderbilt Scale. | 4 & 6 months after enrollment
  We will compare side effects between the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Wasserman, MD, MPH, Principal Investigator — University of Vermont; Alexander G Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- American Academy of Pediatrics, Elk Grove Village, Illinois, United States

REFERENCES:
- See also: ePROS website — http://www.aap.org/